CLINICAL TRIAL: NCT01194141
Title: Safety and Efficacy of Aerobic Exercise Training in Barth Syndrome
Brief Title: Exercise Training in Barth Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, W. Todd Cade, Assisant Professor of Physical Therapy and Medicine, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0652
Record Dates: First submitted 2010-08-30; First posted 2010-09-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Barth Syndrome
Keywords: Barth syndrome; cardiomyopathy; mitochondria; cardiolipin
MeSH Terms: conditions — Barth Syndrome; Cardiomyopathies | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise training (Experimental): Aerobic exercise training 45-60 min/3x/week/12 weeks
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — aerobic exercise training, 45-60 minutes, 3x/week, 12 weeks (3-months)

SUMMARY:
Barth syndrome (BTHS) is a genetic disease that results in heart failure, muscle weakness and exercise intolerance. Several studies in non-BTHS heart failure suggest that endurance exercise training is beneficial in improving exercise intolerance, heart function and quality of life in young men with BTHS. This study will examine the effects of Endurance (i.e. aerobic) exercise training on exercise tolerance, heart function, and quality of life in adolescents and young adults with BTHS. We hypothesize that 3 months of endurance training will improve exercise tolerance, heart function and quality of life in adolescents and young men with BTHS.

DETAILED DESCRIPTION:
Barth Syndrome (BTHS) is an X-linked disorder characterized by severe mitochondrial dysfunction, skeletal and cardiomyopathy and growth retardation. The investigators have recently found severe exercise intolerance in adolescents with BTHS that was mediated by impaired skeletal muscle oxygen extraction and utilization. Previous evidence from other mitochondrial pathologies demonstrated that chronic aerobic exercise training enhanced mitochondrial biogenesis, improved skeletal muscle oxygen extraction/utilization, exercise tolerance and quality of life in these individuals. Chronic aerobic exercise training also improved left ventricular and cardio-autonomic function and decreased the occurrence of arrhythmias in non-Barth heart failure and arrhythmia human and animal models. Currently it is unknown if chronic aerobic exercise training is effective in improving left ventricular function, skeletal muscle mitochondrial biogenesis and oxygen extraction/utilization, exercise tolerance, cardio-autonomic function and quality of life in those with BTHS; a condition containing characteristics consistent with both mitochondrial myopathy and heart failure. Establishing the safety and efficacy of aerobic exercise training in BTHS could lead to clinical recommendations of regular exercise training for the standard of care treatment of individuals with BTHS. It may also provide novel mechanistic information about the adaptability of muscle mitochondria in BTHS. Therefore, the overall objective of the pilot/feasibility/proof-of-concept proposal is to collect preliminary data on the following hypothesis: Supervised aerobic exercise training (3x/wk, 20-45 min, 12 wks) will improve skeletal muscle oxygen extraction/utilization, left ventricular function, peak exercise tolerance, cardio-autonomic function and quality of life, and will be found safe in adolescents and young adults with BTHS. The investigators aim to address these hypotheses through left ventricular function, skeletal muscle oxygen extraction/utilization, and whole body oxygen consumption measurements during a graded exercise test at baseline and following a 3 month supervised aerobic exercise training program in 5 BTHS patients (ages 15-30 yrs). Cardio-autonomic function will be examined using post-exercise heart rate recovery measurements obtained at baseline and after the 12 wk intervention. Supervised exercise training programs will be uniformly designed, but individualized and performed at a hospital based physical therapy or cardiac rehabilitation facility near the participant's home. Left ventricular function will be examined using 2-D, Doppler and Tissue Doppler echocardiography, skeletal muscle oxygen extraction/utilization will be measured using near infrared spectroscopy, whole body oxygen consumption will be measured using indirect calorimetry, cardio-autonomic function will be measured using electrocardiography and quality of life will be measured by the Minnesota Living with Heart Failure Questionnaire (MLWHFQ). The investigators expect to find that exercise training is safe in BTHS, and effectively improves cardiac and skeletal muscle function and quality of life. Preliminary data from this proposal will be used in larger federal or association grant applications examining the cardiovascular, musculo-skeletal and autonomic effects of chronic aerobic exercise training in BTHS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-30 years
2. Sedentary (exercises less than 2x/wk)
3. Motivated to exercise
4. Stable on medications for ≥ 3 months
5. Lives in North America.
6. Planning on attending the Barth Syndrome International Conference in July 2010.

Exclusion Criteria:

1. Unstable heart disease
2. Any concurrent disease that may contraindicate exercise testing and training.
3. Cardiac transplantation

Ages: 15 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption | Enrollment and 3 months
  peak oxygen consumption measured by indirect calorimetry

SECONDARY OUTCOMES:
Cardiac output | Enrollment and 3 months
  cardiac output measured by echocardiography
muscle oxygen extraction | Enrollment and 3 months
  skeletal muscle oxygen extraction measured by near infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: William T Cade, PT, PhD, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Result] Cade WT, Reeds DN, Peterson LR, Bohnert KL, Tinius RA, Benni PB, Byrne BJ, Taylor CL. Endurance Exercise Training in Young Adults with Barth Syndrome: A Pilot Study. JIMD Rep. 2017;32:15-24. doi: 10.1007/8904_2016_553. Epub 2016 Jun 11. PMID 27295193
- See also: Related Info — http://www.barthsyndrome.org